## Informed consent

## A Multicenter Prospective Cohort Study On The Risk Factors for Gallbladder Cancer

Researcher: Wang Jianming

Research Institute: Huazhong University of Science

Tongji Hospital, Tongji Medical College

Date: August 31, 2018

## Informed consent

Patient's cosent for the publication of material relating to them in domestic and international academic journals.

**Clinical Research Project Name:** A Multicenter Prospective Cohort Study of Risk Factors for Gallbladder Cancer **Research Institute:** Huazhong University of Science Tongji Hospital, Tongji Medical College Name: (Name Of Person Described In Article Or Shown In Photograph ) I give my consent for this material to appear in academic journals and associated publications. I have seen any pictures and read the material to be published. I understand that: My name will not be published. I understand, however, that complete anonymity cannot guaranteed. The material may be published and placed on worldwide website and journals. Both the printed version and the website are seen and read by doctors, journalists, and members of the public. The material will not be used for advertising or packaging. I understand that such imaging records may be used for the purpose of informing the medical profession or the general public about characteristics of galbladder cancer, surgery methods, results, issues, trends, concerns and similar maters. Parent/Guardian Date

Witness/physician